CLINICAL TRIAL: NCT05789004
Title: Efficacy of Tooth Bleaching With 35% and 6% Hydrogen Peroxide in Primary Dentition: Study Protocol for a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Tooth Bleaching With 35% and 6% Hydrogen Peroxide in Primary Dentition
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DeciduousBleaching
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Sensitivity, Tooth
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tooth Bleaching

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen Peroxide 35% (Experimental): In the participants of this group, the tooth whitening process will be performed with 35% hydrogen peroxide.
  Interventions: Procedure: Tooth Bleaching with Whiteness HP Automixx 35%
- Hydrogen Peroxide 6% (Experimental): In the participants of this group, the tooth whitening process will be performed with 6% hydrogen peroxide.
  Interventions: Procedure: Tooth Bleaching with Whiteness HP Automixx 6%

INTERVENTIONS:
Procedure: Tooth Bleaching with Whiteness HP Automixx 35% — * Clinical examination and taking the initial shade of the tooth with Vita Easyshade®;
  * Sensitivity/pain recording using the Pain Level Scale (Wong-Baker Faces®);
  * Prophylaxis with a Robson brush and prophylactic paste;
  * Application of lip balm on the patient's lips;
  * Placement of the labial retractor;
  * Application of the gingival barrier;
  * Application of Whiteness HP Automixx 35% whitening gel;
  * In the session, a single application of the gel will be carried out and where it will remain on the surface of the tooth for 15 min;
  * The gel must be removed from the teeth with a sucker and the teeth cleaned with gauze;
  * Sensitivity/pain recording using the Pain Level Scale (Wong-Baker Faces®);
  * The second bleaching session will be carried out 7 days after the first one and, if necessary, a third session can be carried out 7 days after the second one.
  Arms: Hydrogen Peroxide 35%
Procedure: Tooth Bleaching with Whiteness HP Automixx 6% — * Clinical examination and taking the initial shade of the tooth with Vita Easyshade®;
  * Sensitivity/pain recording using the Pain Level Scale (Wong-Baker Faces®);
  * Prophylaxis with a Robson brush and prophylactic paste;
  * Application of lip balm on the patient's lips;
  * Placement of the labial retractor;
  * Application of the gingival barrier;
  * Application of Whiteness HP Automixx 6% whitening gel;
  * In the session, a single application of the gel will be carried out and where it will remain on the surface of the tooth for 15 min;
  * The gel must be removed from the teeth with a sucker and the teeth cleaned with gauze;
  * Sensitivity/pain recording using the Pain Level Scale (Wong-Baker Faces®);
  * The second bleaching session will be carried out 7 days after the first one and, if necessary, a third session can be carried out 7 days after the second one.
  Arms: Hydrogen Peroxide 6%

SUMMARY:
The aesthetics of dental elements generates great psychological and social impacts, both in the deciduous and permanent dentition. One of the techniques widely used to visually improve the appearance of teeth is bleaching. Bleaching can be performed both at home and in a dental office. In office whitening, the technique used consists of applying the whitening gel to the dental surfaces in concentrations ranging from 25% to 50% of hydrogen peroxide. However, recent studies show that low and medium concentration bleaching agents based on hydrogen peroxide have been effective and present a lower risk of sensitivity to the patient. In view of the above, this study aims to carry out a controlled and randomized clinical trial to compare the effectiveness of dental bleaching in deciduous teeth with hydrogen peroxide at concentrations of 35% and 6%. For this, 38 patients aged 03 to 06 years will be selected, allocated in 2 groups (G1 - Hydrogen Peroxide 35%, n=19 and G2- Hydrogen Peroxide 6%, n=19). Bleaching will be carried out in up to three sessions, with an interval of 7 days between them and the evaluation of color and tooth sensitivity will be carried out 48 hours after each bleaching session. The color assessment will be measured using a digital spectrometer and tooth sensitivity using the Pain Level Scale (Wong-Baker Faces®). Descriptive statistical analysis will be carried out, containing the mean and standard deviation in the calculation and normality and homogeneity tests will be carried out, for subsequent adequate statistical analysis. As a result, it is expected that there is no significant difference between the groups in terms of color variation and that the low-concentration bleaching group has the lowest sensitivity index.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 03 to 06 years old;
* Vital or non-vital teeth (already endodontically treated) with severe to moderate discoloration;
* No active carious lesions;
* No lesions in the oral cavity;
* No report of previous tooth sensitivity.

Exclusion Criteria:

- Patients who during anamnesis report allergies to dyes or latex, who withdraw from participating in the study, as well as those who do not attend the callbacks, will be excluded.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Changes in tooth color | Baseline and 48 hours after each bleaching session.
  The Vita Easyshade® digital spectrometer (VITA Zahnfabrik H. Rauter GmbH & Co. KG, Germany) will be used for evaluation. The upper left canine will be used as a color reference because it is the most saturated tooth in the arch (greater dentin mass and greater amount of intrinsic pigments).
Changes in tooth sensitivity | Baseline and 48 hours after each bleaching session.
  It will be explained to the participant that each face drawn in a figure represents a person who has no pain, or some, or a lot of pain. Face 0 doesn't hurt at all. Face 2 hurts a little. Face 4 hurts a little more. Face 6 hurts a lot. Face 8 hurts the most. Face 10 hurts as much as you can imagine, although you don't have to be crying to have this worst pain. The participant will choose the face that best portrays the pain they are experiencing.